CLINICAL TRIAL: NCT05921903
Title: A Phase 2b, Randomized, Controlled, Open-label Study to Evaluate the Immune Response and Safety of the RSVPreF3 OA Investigational Vaccine in Adults (>=18 Years of Age) When Administered to Lung and Renal Transplant Recipients Comparing 1 Versus 2 Doses and Compared to Healthy Controls (>=50 Years of Age) Receiving 1 Dose.
Brief Title: A Study on the Immune Response and Safety of an RSV Vaccine When Given to Adults 18 Years of Age and Above Who Received Lung or Kidney Transplant and Are at an Increased Risk of Respiratory Syncytial Virus Lower Respiratory Tract Disease and Compared to Healthy Adults 50 Years of Age and Above
Acronym: RSV OA=ADJ-023
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 219900; 2023-503951-81-00 (Other: EU CT number)
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Vaccine; Immunogenicity; Safety
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: This study is an open label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- RSV_IC_1 group (Experimental): Immunocompromised (IC) participants (recipients of lung or renal transplant) received 1 dose of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1).
  Interventions: Biological: RSVPreF3 OA Investigational Vaccine
- RSV_IC_2 group (Experimental): IC participants (recipients of lung or renal transplant) received 2 doses of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1) and Visit 3 (Visit 1 + 30-60 days).
  Interventions: Biological: RSVPreF3 OA Investigational Vaccine
- RSV_HA group (Active Comparator): Healthy adult (HA) participants received 1 dose of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1).
  Interventions: Biological: RSVPreF3 OA Investigational Vaccine

INTERVENTIONS:
Biological: RSVPreF3 OA Investigational Vaccine — 0.5 mililiter dose was administered intramuscularly as 1 dose to RSV_IC_1 and RSV_HA groups, and 2 doses to RSV_IC_2 group.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity, safety, and reactogenicity of the RSVPreF3 OA investigational vaccine in an immunocompromised (lung and renal transplant recipients) population and assess whether a second dose of the vaccine increases the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Participants and/or participant's parent(s)/LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance can be enrolled, such that the participant is primarily responsible for self-care and activities of daily living.
* Written or witnessed informed consent obtained from the participant/participant's parent(s)/LAR(s) (participant must be able to understand the informed consent) prior to performance of any study-specific procedure.
* Female participants of nonchildbearing potential may be enrolled in the study. Non-childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, and post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant has practiced adequate contraception from 1 month prior to study intervention administration and agreed to continue adequate contraception until study end for this study, and has a negative pregnancy test on the day of and prior to study intervention administration.

Specific inclusion criteria for renal/lung transplant patients:

* A male or female, >=18 YoA at the time of signing the Informed consent form (ICF) or Informed assent form (IAF).
* Written informed assent obtained from the participant (participant must be able to understand the informed assent) if he/she is less than legal age of consent, or written informed consent obtained from the participant if the participant has achieved legal age of consent.
* Participant who has received an ABO compatible allogeneic renal or lung transplant (allograft) more than 12 months (365 days) prior to the first study intervention administration.
* Participant receiving maintenance immunosuppressive therapy for the prevention of allograft rejection.

Specific inclusion criteria for renal transplant (RTx) patients:

• Participant with stable renal function, stability defined as less than 20% variability between last two results of eGFR or in the opinion of the investigator after investigator review of more than the last two results of eGFRs and based on medical history.

Specific inclusion criteria for lung transplant (LTx) patients:

• Participant with stable lung function, with stability defined as the stability in the FEV1 compared to post-transplant baseline FEV1 and based on medical history of the last 3 months, in the opinion of the investigator.

Specific inclusion criteria for healthy participants:

* A male or female, >=50 YoA at the time of signing the ICF.
* Healthy participants as established by medical history and clinical examination before entering the study.
* Participants who are medically stable in the opinion of the investigator at the time of first study intervention administration.
* Participants with chronic stable medical conditions with or without specific treatment, such as diabetes mellitus, hypertension, or cardiac disease, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

Medical conditions:

* History of any reaction/ hypersensitivity likely to be exacerbated by any component of the study intervention.
* Acute or chronic clinically significant cardiovascular or hepatic functional abnormality as determined by physical examination or laboratory screening tests.
* Recurrent/uncontrolled neurological disorders or seizures. Participants with medically controlled chronic neurological diseases can be enrolled in the study if their condition will allow them to comply with the requirements of the protocol, with the help of a caregiver if needed.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Any condition which would make IM injection unsafe.
* Significant underlying illness that would prevent completion of the study).
* Acute disease and/or fever at the time of study intervention administration (>=38°C /100.4°F, oral or axillary). Participants with a minor illness without fever may be enrolled at the discretion of the investigator.
* Bedridden participants.

Prior/Concomitant therapy:

* Use of any other investigational or non-registered product (drug, vaccine, or medical device) up to 30 days before the first dose administration (Day -30 to Day 1), or their planned use during the study period (up to Visit 6).
* Previous vaccination with the study antigen (RSV), including investigational RSV vaccines.
* Unexpected vaccine administration during a study should not occur 30 days prior to the first dose or 30 days after the last dose. For COVID-19 and inactivated/subunit/split influenza vaccines, this window is shortened to 14 days.

Prior/Concurrent clinical study experience:

• Concurrently participating in another active clinical study

Other exclusion criteria:

* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse
* Participation of any study personnel or their immediate dependents.
* Planned move during the study period that will prohibit participating in the study until study end.

Specific exclusion criteria for renal/lung transplant patients:

* More than one organ transplanted. Dual organ is allowed.
* History of events that may put the participant at increased risk for chronic allograft dysfunction.
* Participant with an episode of allograft rejection over the previous 90 days prior to the first study intervention administration.
* Histologic evidence of chronic allograft injury.
* Active treatment for acute rejection.
* Current diagnosis of malignancy (except non-melanoma skin cancer that does not require systemic therapy).
* Any autoimmune conditions or pIMDs that may put the participant at increased risk.
* Any confirmed or suspected HIV infection, primary immunodeficiency disease or ongoing CMV infection with a viremia >200 IU/mL.
* Use of anti-CD20 or other B-cell monoclonal antibody agents for the prevention of allograft rejection within 274 days of first dose of study.
* Use of investigational and non-registered immunosuppressants at the local/country level, unless specifically prescribed for the prevention of allograft rejection, and which are in process of approval, approved in other countries and locally available.
* Evidence/high suspicion\ of noncompliance/nonadherence to use of induction and/or maintenance immunosuppressive therapies.
* Any clinically significant hematologic and/or biochemical laboratory abnormality.

Specific exclusion criteria for RTx patients:

* Previous allograft loss secondary to recurrent primary kidney disease. Multiple consecutive kidney transplants are allowed if the reason is not recurrent primary kidney disease.
* Evidence of significant proteinuria/albuminuria.

Specific exclusion criteria for LTx patients:

* At study intervention administration visit, diagnosis of documented acute pulmonary infection within the 2 prior weeks.
* Patients with diagnosis of chronic lung allograft dysfunction (decrement of >=20% in FEV1 compared to post-transplant baseline FEV1).

Specific exclusion criteria for healthy participants:

* Any confirmed/suspected immunosuppressive/immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination.
* Unstable serious chronic illness.
* Chronic administration of immune-modifying drugs (>14 days in total) and/or administration of long-acting immune-modifying treatments or planned administration at any time up to the end of the study.

  * Up to 3 months prior to the study intervention administration:
  * For corticosteroids -prednisone equivalent ≥20 mg/day, or equivalent. Inhaled, topical and intra-articular steroids are allowed.
  * Administration of immunoglobulins and/or any blood products or plasma derivatives.
  * Up to 6 months prior to study intervention administration: long-acting immune-modifying drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2025-05-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (9):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Temple, Texas
- Australia (4):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Birtinya, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Adelaide, South Australia
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec
- GSK Investigational Site, Giessen, Germany
- Italy (4):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Siena
- Japan (6):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Derived] Vyse A, Hockey C, Wright H, Ellsbury G. Could more adults than just those aged 75-79 years potentially benefit from vaccination against RSV: insights from UK data. J Pharm Policy Pract. 2025 Nov 4;18(1):2576618. doi: 10.1080/20523211.2025.2576618. eCollection 2025. PMID 41199924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from 48 study sites were enrolled in the study.
Pre-assignment Details: All participants enrolled were randomized to the Exposed set and started the study. Analysis presented includes data up to Primary Completion. Additional results will be provided within one year of study completion.
Period: Overall Study
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Started | 131 | 130 | 125
Completed | 2 | 0 | 12
Not Completed | 129 | 130 | 113
Not completed — Unsolicited non-SAE | 0 | 1 | 0
Not completed — SAEs/pIMDs/AESIs specific to SOT | 0 | 3 | 1
Not completed — Ongoing at the time of Primary Completion Analysis | 129 | 126 | 112

BASELINE CHARACTERISTICS:
Population: Exposed set included all participants that received at least one study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group | Total
Number analyzed (Participants) | 131 | 130 | 125 | 386
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 61.9 (9.3) | 61.4 (8.4) | 63.8 (8.2) | 62.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 50 | 66 | 170
  Male | 77 | 80 | 59 | 216
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Races where 0<n<11 (i.e., ASIAN, AMERICAN INDIAN OR ALASKA NATIVE, BLACK OR AFRICAN AMERICAN, NOT REPORTED, MULTIPLE and UNKNOWN) are combined into one category ("All Other Races") to maintain participant confidentiality and privacy.
  Participants
    White | 89 | 79 | 95 | 263
    All Other Races | 42 | 51 | 30 | 123

OUTCOME MEASURES:

1. Primary Outcome: RSV-A Serum Neutralizing Titers Expressed As Mean Geometric Increase (MGI) Post-Dose 2 (Visit 4) Over Post-Dose 1 (Visit 3) for RSV_IC_2 Group
Description: MGI was defined as the geometric mean of the within-participant ratios of serum neutralizing titers against RSV-A post-Dose 2 (Visit 4) over post-Dose 1 (Visit 3).
Time Frame: At Visit 4 (Visit 3 + 30-42 days) compared with Visit 3 (Visit 1 [Day 1] + 30-60 days)
Population: Analysis was performed on the Per protocol Set (PPS) for humoral immunogenicity, which included all participants who received the study intervention administration as per protocol, had immunogenicity results pre and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity, without prohibited concomitant medication/vaccination. Only participants with data available at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RSV_IC_2 Group
Number analyzed (Participants) | 111
Ratio | 1.34 [1.20 to 1.48]

2. Primary Outcome: RSV-B Serum Neutralizing Titers Expressed As MGI Post-Dose 2 (Visit 4) Over Post-Dose 1 (Visit 3) for RSV_IC_2 Group
Description: MGI was defined as the geometric mean of the within-participant ratios of serum neutralizing titers against RSV-B post-Dose 2 (Visit 4) over post-Dose 1 (Visit 3).
Time Frame: At Visit 4 (Visit 3 + 30-42 days) compared with Visit 3 (Visit 1 [Day 1] + 30-60 days)
Population: Analysis was performed on PPS for humoral immunogenicity. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | RSV_IC_2 Group
Number analyzed (Participants) | 111
Ratio | 1.26 [1.14 to 1.40]

3. Secondary Outcome: RSV-A And RSV-B Serum Neutralizing Titers Expressed As Geometric Mean Titers (GMT) for RSV_IC_1, RSV_IC_2 and RSV_HA Groups
Description: Neutralizing titers were calculated as GMT and expressed in titers (Estimated Dilution 60 [ED60]).
Time Frame: At pre-study intervention administration (at Visit 1 [Day 1]), Visit 2 in a subset of participants (Visit 1 + 7-14 days), Visit 3 (Visit 1 + 30-60 days) and Visit 4 (Visit 3 + 30-42 days)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Groups:
- RSV_HA Group: Healthy participants received 1 dose of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1).
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 123 | 123 | 125
Titers (ED60)
  RSV-A , Visit 1 | 807.0 [700.9 to 929.2] | 814.1 [701.3 to 945.1] | 889.0 [781.9 to 1010.6]
  RSV-A , Visit 2: number analyzed (Participants) | 36 | 36 | 34
  RSV-A , Visit 2 | 1775.8 [1201.0 to 2625.6] | 2031.1 [1283.6 to 3213.9] | 6716.8 [4907.6 to 9193.0]
  RSV-A , Visit 3: number analyzed (Participants) | 123 | 114 | 118
  RSV-A , Visit 3 | 3990.8 [3219.4 to 4947.0] | 4174.0 [3230.7 to 5392.6] | 6822.5 [5926.2 to 7854.4]
  RSV-A , Visit 4: number analyzed (Participants) | 116 | 111 | 110
  RSV-A , Visit 4 | 4184.7 [3360.1 to 5211.7] | 5377.9 [4265.4 to 6780.6] | 5707.0 [4853.6 to 6710.3]
  RSV-B, Visit 1 | 864.2 [727.8 to 1026.2] | 892.9 [754.1 to 1057.3] | 1027.3 [889.6 to 1186.3]
  RSV-B, Visit 2: number analyzed (Participants) | 36 | 36 | 34
  RSV-B, Visit 2 | 2325.3 [1592.9 to 3394.5] | 2603.1 [1714.9 to 3951.3] | 8113.6 [5699.9 to 11549.5]
  RSV-B, Visit 3: number analyzed (Participants) | 123 | 114 | 118
  RSV-B, Visit 3 | 5002.9 [3901.7 to 6414.8] | 4834.7 [3736.6 to 6255.6] | 9140.5 [7805.3 to 10704.1]
  RSV-B, Visit 4: number analyzed (Participants) | 116 | 111 | 110
  RSV-B, Visit 4 | 4461.7 [3519.0 to 5657.0] | 5820.8 [4658.2 to 7273.5] | 6281.6 [5377.6 to 7337.7]

4. Secondary Outcome: RSV-A and RSV-B Serum Neutralizing Titers Expressed as GMT for RSV_IC_1, RSV_IC_2 and RSV_HA Groups
Description: Neutralizing titers were calculated as GMT and expressed in titers (ED60).
Time Frame: At Visit 5 (last dose + 180-210 days) and Visit 6 (last dose + 350-380 days)
Reporting Status: Not Posted

5. Secondary Outcome: RSV-A Serum Neutralizing Titers Expressed As Group GMT For RSV_HA And Pooled RSV_IC Groups
Description: Group GMT was assessed for RSV_HA group over pooled RSV_IC group (combined RSV_IC_1 and RSV_IC_2 groups). The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_HA and Pooled RSV_IC groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 2 in a subset of participants (Visit 1 [Day 1] + 7-14 days) and Visit 3 (Visit 1 + 30-60 days)
Population: Analysis was performed on PPS for humoral immunogenicity. Only participants with data available for the specified groups at the specified timepoints were included in this analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Groups:
- Pooled RSV_IC Group: IC participants (recipients of lung or renal transplant) who received 1 dose of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1) in RSV_IC_1 and RSV_IC_2 groups were pooled, as pre-specified in the statistical analysis plan for humoral immunogenicity analysis up to Visit 3 (Visit 1 + 30-60 days).
Arm/Group | RSV_HA Group | Pooled RSV_IC Group
Number analyzed (Participants) | 118 | 235
Titers (ED60)
  Visit 2: number analyzed (Participants) | 34 | 72
  Visit 2 | 6689.9 [4639.3 to 9646.7] | 1902.8 [1479.6 to 2446.9]
  Visit 3 | 6653.8 [5503.5 to 8044.6] | 4113.0 [3595.5 to 4705.0]
Statistical Analysis 1: Comparison: RSV_HA Group vs Pooled RSV_IC Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant (Pooled RSV_IC group) and healthy participants (RSV_HA group) for the RSV-A strain at Visit 2; Test type: Other — The statistical analyses performed for the study objectives were descriptive. No success criteria were defined for the statistical analyses conducted in this study; ANCOVA; GMT Ratio = 3.52, 95% CI 2-sided [2.26 to 5.48] — The comparison is done using the group ratio of adjusted GMT (RSV_HA/Pooled RSV_IC) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate
Statistical Analysis 2: Comparison: RSV_HA Group vs Pooled RSV_IC Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant (Pooled RSV_IC group) and healthy participants (RSV_HA group) for the RSV-A strain at Visit 3; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.62, 95% CI 2-sided [1.28 to 2.04] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: RSV-A Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_1 And RSV_IC_2 Groups
Description: Group GMT of RSV_IC_2 over RSV_IC_1 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing titers included the baseline log10-transformed titer and the SOT type as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_1 and RSV_IC_2 groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group
Number analyzed (Participants) | 114 | 110
Titers (ED60) | 4041.9 [3254.8 to 5019.3] | 5098.4 [4088.8 to 6357.3]
Statistical Analysis 1: Comparison: RSV_IC_1 Group vs RSV_IC_2 Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 1 dose of vaccine (RSV_IC_1 group) and participants that received lung or kidney solid organ transplant and 2 doses of vaccine (RSV_IC_2 group) for the RSV-A strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.26, 95% CI 2-sided [0.94 to 1.69] — The comparison is done using the group ratio of adjusted GMT (RSV_IC_2/RSV_IC_1) (ANCOVA model applied to the log10- transformed titers). ANCOVA model included the group as fixed effect, and SOT type and baseline log10-transformed titer as covariate

7. Secondary Outcome: RSV-A Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_1 And RSV_HA Groups
Description: Group GMT of RSV_HA over RSV_IC_1 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_1 and RSV_HA groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_1 Group | RSV_HA Group
Number analyzed (Participants) | 114 | 110
Titers (ED60) | 4244.8 [3551.8 to 5073.0] | 5541.6 [4622.0 to 6644.2]
Statistical Analysis 1: Comparison: RSV_IC_1 Group vs RSV_HA Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 1 dose of study intervention (RSV_IC_1 group) and healthy participants (RSV_HA group) for the RSV-A strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.31, 95% CI 2-sided [1.01 to 1.68] — The comparison is done using the group ratio of adjusted GMT (RSV_HA/RSV_IC_1) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate

8. Secondary Outcome: RSV-A Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_2 And RSV_HA Groups
Description: Group GMT of RSV_HA over RSV_IC_2 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-A neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_2 and RSV_HA groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 110 | 110
Titers (ED60) | 5505.3 [4627.0 to 6550.3] | 5615.7 [4719.8 to 6681.6]
Statistical Analysis 1: Comparison: RSV_IC_2 Group vs RSV_HA Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 2 doses of study intervention (RSV_IC_2 group) and healthy participants (RSV_HA group) for the RSV-A strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.02, 95% CI 2-sided [0.80 to 1.30] — The comparison is done using the group ratio of adjusted GMT (RSV_HA/RSV_IC_2) (ANCOVA model applied to the log10- transformed titers). The ANCOVA model included the group as fixed effects and the pre-dose log-10 titer as covariate

9. Secondary Outcome: RSV-A Serum Neutralizing Titers Expressed as Group GMT for RSV_IC_1, RSV_IC_2 and RSV_HA Groups
Time Frame: At Visit 5 (last dose + 180-210 days) and Visit 6 (last dose + 350-380 days)
Reporting Status: Not Posted

10. Secondary Outcome: RSV-B Serum Neutralizing Titers Expressed As Group GMT For RSV_HA And Pooled RSV_IC Groups
Description: Group GMT was assessed for RSV_HA group over pooled RSV_IC group (combined RSV_IC_1 and RSV_IC_2 groups). The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_HA and Pooled RSV_IC groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 2 in a subset of participants (Visit 1 [Day 1] + 7-14 days) and Visit 3 (Visit 1 + 30-60 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_HA Group | Pooled RSV_IC Group
Number analyzed (Participants) | 118 | 235
Titers (ED60)
  Visit 2: number analyzed (Participants) | 34 | 72
  Visit 2 | 8238.7 [5972.9 to 11364.1] | 2442.6 [1958.3 to 3046.7]
  Visit 3 | 8545.5 [7031.3 to 10385.8] | 5106.9 [4448.4 to 5863.0]
Statistical Analysis 1: Comparison: RSV_HA Group vs Pooled RSV_IC Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant (Pooled RSV_IC group) and healthy participants (RSV_HA group) for the RSV-B strain at Visit 2; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 3.37, 95% CI 2-sided [2.28 to 4.98] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: RSV_HA Group vs Pooled RSV_IC Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant (Pooled RSV_IC group) and healthy participants (RSV_HA group) for the RSV-B strain at Visit 3; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.67, 95% CI 2-sided [1.32 to 2.13] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: RSV-B Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_1 And RSV_IC_2 Groups
Description: Group GMT ratio of RSV_IC_2 over RSV_IC_1 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing titers included the baseline log10-transformed titer and the SOT type as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_1 and RSV_IC_2 groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group
Number analyzed (Participants) | 114 | 110
Titers (ED60) | 4333.3 [3510.0 to 5349.8] | 5550.5 [4478.3 to 6879.4]
Statistical Analysis 1: Comparison: RSV_IC_1 Group vs RSV_IC_2 Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 1 dose of vaccine (RSV_IC_1 group) and participants that received lung or kidney solid organ transplant and 2 doses of vaccine (RSV_IC_2 group) for the RSV-B strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.28, 95% CI 2-sided [0.97 to 1.70] — [estimate comment as in outcome 6, analysis 1]

12. Secondary Outcome: RSV-B Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_1 And RSV_HA Groups
Description: Group GMT of RSV_HA over RSV_IC_1 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_1 and RSV_HA groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_1 Group | RSV_HA Group
Number analyzed (Participants) | 114 | 110
Titers (ED60) | 4632.9 [3890.8 to 5516.6] | 5973.5 [5000.9 to 7135.4]
Statistical Analysis 1: Comparison: RSV_IC_1 Group vs RSV_HA Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 1 dose of study intervention (RSV_IC_1 group) and healthy participants (RSV_HA group) for the RSV-B strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.29, 95% CI 2-sided [1.00 to 1.65] — [estimate comment as in outcome 7, analysis 1]

13. Secondary Outcome: RSV-B Serum Neutralizing Titers Expressed As Group GMT For RSV_IC_2 And RSV_HA Groups
Description: Group GMT of RSV_HA over RSV_IC_2 was assessed at Visit 4. The ANCOVA model used to calculate the adjusted GMTs for RSV-B neutralizing titers included the baseline log10-transformed titer as covariate (i.e. GMTs are adjusted for the PRE timepoint values) and only included RSV_IC_2 and RSV_HA groups in the model as fixed effect, as specified in Statistical Analysis Plan.
Time Frame: At Visit 4 (Visit 3 [Visit 1 (Day 1) + 30-60 days] + 30-42 days)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (ED60)
Arm/Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 110 | 110
Titers (ED60) | 6090.6 [5184.6 to 7155.0] | 6123.0 [5212.1 to 7193.0]
Statistical Analysis 1: Comparison: RSV_IC_2 Group vs RSV_HA Group; To evaluate the humoral immune response to the RSVPreF3 OA investigational vaccine in participants that received lung or kidney solid organ transplant and 2 doses of study intervention (RSV_IC_2 group) and healthy participants (RSV_HA group) for the RSV-B strain at Visit 4; Test type: Other — [test comment as in outcome 5, analysis 1]; ANCOVA; GMT Ratio = 1.01, 95% CI 2-sided [0.80 to 1.26] — [estimate comment as in outcome 8, analysis 1]

14. Secondary Outcome: RSV-B Serum Neutralizing Titers Expressed as Group GMT for RSV_IC_1, RSV_IC_2 and RSV_HA Groups
Time Frame: At Visit 5 (last dose +180-210 days) and Visit 6 (last dose + 350-380 days)
Reporting Status: Not Posted

15. Secondary Outcome: RSV-A And RSV-B Serum Neutralizing Titers Expressed As MGI
Description: MGI was assessed at Visit 2 (in a subset of participants) over Visit 1 and Visit 3 over Visit 1 in RSV_HA and pooled RSV_IC (combined RSV_IC_1 and RSV_IC_2 groups), and at Visit 4 over Visit 1 in RSV_IC_1, RSV_IC_2, RSV_HA groups.
Time Frame: At Visit 2 in a subset of participants (Visit 1 [Day 1] + 7-14 days), Visit 3 (Visit 1 + 30-60 days) and Visit 4 (Visit 3 + 30-42 days), each compared to Visit 1 (Day 1)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Pooled RSV_IC Group: IC participants (recipients of lung or renal transplant) who received 1 dose of RSVPreF3 OA investigational vaccine at Visit 1 (Day 1) in RSV_IC_1 and RSV_IC_2 groups were pooled. As pre-specified in the statistical analysis plan, the IC participants were pooled for humoral immunogenicity analysis up to Visit 3 (Visit 1 + 30-60 days).
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group | Pooled RSV_IC Group
Number analyzed (Participants) | 122 | 113 | 118 | 235
Ratio
  RSV-A, Visit 2: number analyzed (Participants) | 36 | 36 | 34 | 72
  RSV-A, Visit 2 | 2.14 [1.44 to 3.18] | 2.20 [1.45 to 3.34] | 7.59 [5.44 to 10.58] | 2.17 [1.64 to 2.87]
  RSV-A, Visit 3 | 4.92 [3.95 to 6.12] | 5.01 [4.00 to 6.27] | 7.82 [6.74 to 9.06] | 4.96 [4.24 to 5.80]
  RSV-A, Visit 4: number analyzed (Participants) | 114 | 110 | 110 | 0
  RSV-A, Visit 4 | 5.29 [4.24 to 6.60] | 6.53 [5.32 to 8.01] | 6.55 [5.60 to 7.6] |
  RSV-B, Visit 2: number analyzed (Participants) | 36 | 36 | 34 | 72
  RSV-B, Visit 2 | 2.51 [1.78 to 3.55] | 2.54 [1.75 to 3.67] | 8.59 [6.59 to 11.20] | 2.53 [1.98 to 3.23]
  RSV-B, Visit 3 | 5.72 [4.53 to 7.21] | 5.34 [4.25 to 6.72] | 8.80 [7.67 to 10.11] | 5.53 [4.71 to 6.51]
  RSV-B, Visit 4: number analyzed (Participants) | 114 | 110 | 110 | 0
  RSV-B, Visit 4 | 5.22 [4.20 to 6.49] | 6.52 [5.34 to 7.97] | 6.35 [5.50 to 7.33] |

16. Secondary Outcome: RSV-A and RSV-B Serum Neutralizing Titers Expressed as MGI
Time Frame: At Visit 5 (last dose +180-210 days) and Visit 6 (last dose + 350-380 days), each compared with Visit 1 (Day 1)
Reporting Status: Not Posted

17. Secondary Outcome: Cell Mediated Immunity (CMI) Response In A Subset of Participants Expressed As Group Geometric Mean Of The Frequency Of RSVPreF3-Specific Cluster Of Differentiation (CD) 4+ T Cells
Description: CMI response is expressed as group geometric mean of the frequency of RSVPreF3-specific cluster of differentiation CD4+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-alpha, IFN-gamma, IL- 13 and IL-17. The CMI is measured in a subgroup consisting of participants with renal and lung SOT (from RSV_IC_1 and RSV_IC_2 groups) and healthy participants (from RSV_HA group).
Time Frame: At pre-study intervention administration (at Visit 1 [Day 1]), Visit 2 (Visit 1 + 7-14 days), Visit 3 (Visit 1 + 30-60 days) and Visit 4 (Visit 3 + 30-42 days)
Population: Analysis was performed on the PPS for cell mediated immunity (CMI), which included all participants who received the study intervention administration as per protocol, had cell mediated immunogenicity results pre and post-dose, complied with blood draw intervals, without intercurrent conditions that may interfere with immunogenicity, without prohibited concomitant medication/vaccination. Only participants with data available for CD4+ T cells at the specified timepoints were included in analysis.
Measure: Geometric Mean (Standard Deviation); unit: Specific CD4+ Tcells/million CD4+ Tcells
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 24 | 28 | 31
Specific CD4+ Tcells/million CD4+ Tcells
  Visit 1: number analyzed (Participants) | 23 | 28 | 31
  Visit 1 | 86.8 (1.0) | 110.3 (0.9) | 107.8 (0.9)
  Visit 2: number analyzed (Participants) | 24 | 27 | 28
  Visit 2 | 2932.2 (0.6) | 3704.3 (0.5) | 2959.8 (0.3)
  Visit 3: number analyzed (Participants) | 22 | 28 | 24
  Visit 3 | 1049.0 (0.8) | 1718.5 (0.4) | 1042.4 (0.3)
  Visit 4: number analyzed (Participants) | 23 | 26 | 28
  Visit 4 | 910.8 (0.8) | 2709.0 (0.3) | 734.4 (0.3)

18. Secondary Outcome: CMI Response In A Subset of Participants Expressed As Group Geometric Mean Of The Frequency Of RSVPreF3-Specific CD8+ T Cells
Description: CMI response is expressed as group geometric mean of the frequency of RSVPreF3-specific CD8+ T cells expressing at least 2 activation markers including at least one cytokine among CD40L, 4-1BB, IL-2, TNF-alpha, IFN-gamma, IL- 13 and IL-17. The CMI is measured in a subgroup consisting of participants with renal and lung SOT (from RSV_IC_1 and RSV_IC_2 groups) and healthy participants (from RSV_HA group).
Time Frame: as for outcome 17
Population: Analysis was performed on PPS for CMI. Only participants with data available for CD8+ T cells for the specified groups at the specified timepoints were included in this analysis.
Measure: Geometric Mean (Standard Deviation); unit: Specific CD8+ Tcells/million CD8+ Tcells
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 22 | 25 | 27
Specific CD8+ Tcells/million CD8+ Tcells
  Visit 1: number analyzed (Participants) | 20 | 24 | 27
  Visit 1 | 33.9 (1.0) | 8.2 (1.1) | 27.7 (1.0)
  Visit 2: number analyzed (Participants) | 20 | 23 | 23
  Visit 2 | 16.0 (1.2) | 8.7 (1.0) | 13.0 (1.2)
  Visit 3: number analyzed (Participants) | 20 | 23 | 21
  Visit 3 | 21.7 (0.8) | 22.3 (1.1) | 21.0 (1.1)
  Visit 4: number analyzed (Participants) | 22 | 25 | 24
  Visit 4 | 12.0 (1.1) | 16.9 (0.9) | 13.2 (1.1)

19. Secondary Outcome: CMI Response in a Subset of Participants
Time Frame: At Visit 5 (last dose + 180-210 days) and Visit 6 (last dose + 350-380 days)
Reporting Status: Not Posted

20. Secondary Outcome: Number Of Participants Reporting Any Solicited Administration Site Events
Description: Assessed solicited administration site events included pain, erythema (redness) and swelling, at the injection site. Any = occurrence of the symptom regardless of intensity grade or relation to study intervention.
Time Frame: Within 7 days (i.e., the day of vaccination and 6 subsequent days) after vaccine administration (vaccine administered at Visit 1 [Day 1] for all groups, and Visit 3 [Visit 1 +30-60 days] for RSV_IC_2 group)
Population: Analysis was performed on the Exposed set (ES) which included all participants who received the study intervention administration. Only participants with solicited administration site events at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 131 | 128 | 125
Participants
  Pain, Dosing at visit 1 | 95 | 92 | 95
  Pain, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Pain, Dosing at visit 3 |  | 81 |
  Erythema, Dosing at visit 1 | 8 | 14 | 11
  Erythema, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Erythema, Dosing at visit 3 |  | 10 |
  Swelling, Dosing at visit 1 | 8 | 11 | 3
  Swelling, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Swelling, Dosing at visit 3 |  | 6 |

21. Secondary Outcome: Number Of Participants Reporting Any Solicited Systemic Events
Description: Assessed solicited systemic events included fever (pyrexia), myalgia, arthralgia, headache, and fatigue. Fever is defined as body temperature greater or equal to (≥) 38 degrees Celsius (ºC). Any = occurrence of the symptom regardless of intensity grade or relation to study intervention.
Time Frame: as for outcome 20
Population: Analysis was performed on the ES. Only participants with solicited systemic events at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 131 | 128 | 125
Participants
  Fever , Dosing at visit 1 | 2 | 1 | 1
  Fever , Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Fever , Dosing at visit 3 |  | 2 |
  Myalgia, Dosing at visit 1 | 37 | 38 | 49
  Myalgia, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Myalgia, Dosing at visit 3 |  | 38 |
  Arthralgia, Dosing at visit 1 | 19 | 15 | 15
  Arthralgia, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Arthralgia, Dosing at visit 3 |  | 19 |
  Headache, Dosing at visit 1 | 31 | 33 | 44
  Headache, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Headache, Dosing at visit 3 |  | 30 |
  Fatigue, Dosing at visit 1 | 41 | 45 | 48
  Fatigue, Dosing at visit 3: number analyzed (Participants) | 0 | 118 | 0
  Fatigue, Dosing at visit 3 |  | 47 |

22. Secondary Outcome: Number Of Participants Reporting Any Unsolicited Adverse Events (AEs) At Any Dose Administration
Description: An unsolicited AE is an AE that was not included in the list of solicited events. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is to be reported as an unsolicited AE. Any = occurrence of the symptom regardless of intensity grade or relation to study intervention.
Time Frame: Within 30 days (i.e., the day of vaccination and 29 subsequent days) after vaccine administration (vaccine administered at Visit 1 [Day 1] for all groups, and Visit 3 [Visit 1 +30-60 days] for RSV_IC_2 group)
Population: Analysis was performed on the ES. Only participants with unsolicited AEs at the specified timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 131 | 130 | 125
Participants | 21 | 60 | 26

23. Secondary Outcome: Number Of Participants Reporting Any Serious Adverse Events (SAEs), SAEs Related To Study Intervention And Fatal SAEs
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study participant. Any SAE = occurrence of the SAE regardless of relation to study vaccination. Related SAE = SAE assessed by the investigator as related to the study vaccination. Fatal SAE = occurrence of a fatal SAE regardless of relation to study vaccination.
Time Frame: From Visit 1 (Day 1) up to Visit 4 (Visit 3 + 30-42 days) after vaccine administration (vaccine administered at Visit 1 [Day 1] for all groups, and Visit 3 [Visit 1 + 30-60 days] for RSV_IC_2 group)
Population: Analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 131 | 130 | 125
Participants
  Any SAEs | 12 | 18 | 3
  Related SAEs | 1 | 0 | 0
  Fatal SAEs | 0 | 2 | 0

24. Secondary Outcome: Number Of Participants Reporting Any Potential Immune-Mediated Disease (pIMDs) And pIMDs Related To Study Intervention
Description: pIMDs are a subset of AESIs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any pIMDs = occurrence of the pIMDs regardless of relation to study vaccination. Related pIMDs = pIMDs assessed by the investigator as related to the study vaccination.
Time Frame: as for outcome 23
Population: Analysis was performed on the ES.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
Number analyzed (Participants) | 131 | 130 | 125
Participants
  Any pIMD | 0 | 0 | 1
  Related pIMD | 0 | 0 | 0

25. Secondary Outcome: Number Of Participants With Any AEs Of Special Interest (AESIs) Specific To Renal And Lung SOT Participants
Description: AESIs include the acute rejection of transplant (specific to renal and lung SOT participants). Analysis was performed only on participants that received transplant in RSV_IC_1 and RSV_IC_2 groups.
Time Frame: as for outcome 23
Population: Analysis was performed on the ES. Only SOT participants that had data available at the specified timepoints were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group
Number analyzed (Participants) | 131 | 130
Participants | 0 | 1

26. Secondary Outcome: Number of Participants Reporting Any SAEs, SAEs Related to Study Intervention and Fatal SAEs
Description: as for outcome 23
Time Frame: From Visit 1 (Day 1) up to study end (Visit 6 - last dose + 350-380 days), vaccine administered at Visit 1 [Day 1] for all groups, and Visit 3 [Visit 1 + 30-60 days] for RSV_IC_2 group)
Reporting Status: Not Posted

27. Secondary Outcome: Number of Participants Reporting Any pIMDs and pIMDs Related to Study Intervention
Description: as for outcome 24
Time Frame: as for outcome 26
Reporting Status: Not Posted

28. Secondary Outcome: Number of Participants Reporting Any AESIs Specific to Renal and Lung SOT Participants
Description: as for outcome 25
Time Frame: as for outcome 26
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 7 days post each dose administration, and unsolicited AEs: within 30 days post each dose administration, where doses were administered at Visit 1 [Day 1] for all groups, and Visit 3 [Visit 1(Day 1) + 30-60 days] for RSV_IC_2 group). SAEs, related SAEs, fatal SAEs, pIMDs, related pIMDs and AESIs specific for renal/lung transplant: Visit 1 (Day 1) to Visit 4 (Visit 3 + 30-42 days).
Description: Solicited and unsolicited events were reported per participant at any dose for the assessed timeframe according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | RSV_IC_1 Group | RSV_IC_2 Group | RSV_HA Group
All-Cause Mortality (participants affected / at risk) | 0/131 | 2/130 | 0/125
Serious Adverse Events (participants affected / at risk) | 12/131 | 18/130 | 3/125
Other Adverse Events (participants affected / at risk) | 106/131 | 120/130 | 111/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_IC_1 Group (N=131) | RSV_IC_2 Group (N=130) | RSV_HA Group (N=125)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome with excess blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_IC_1 Group (N=131) | RSV_IC_2 Group (N=130) | RSV_HA Group (N=125)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (4) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymph gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stenotrophomonas maltophilia pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 2 (2) | 1 (1)
Administration site pruritus (General disorders) | 0 (0) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0)
Administration site pain (General disorders) | 95 (95) | 108 (173) | 95 (96)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 41 (41) | 61 (92) | 49 (49)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 32 (32) | 46 (67) | 44 (47)
Dizziness (Nervous system disorders) | 1 (1) | 5 (6) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain fog (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (38) | 56 (77) | 49 (50)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (19) | 27 (36) | 15 (15)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (5) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal mucosal hypertrophy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Administration site erythema (General disorders) | 8 (8) | 19 (24) | 11 (11)
Administration site swelling (General disorders) | 8 (8) | 14 (17) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT05921903/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT05921903/SAP_001.pdf